CLINICAL TRIAL: NCT02349139
Title: A Phase 1/2, Open-Label, Uncontrolled, Multiple-Dose Escalation, Cohort Expansion And Extension Study To Evaluate The Safety, Tolerability, And Pharmacokinetics Of ASN001 In Subjects With Metastatic Progressive Castrate Resistant Prostate Cancer
Brief Title: Safety, Preliminary Efficacy and Pharmacokinetics of ASN001 in Metastatic Castrate Resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Asana BioSciences (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ASN001-101
Record Dates: First submitted 2015-01-13; First posted 2015-01-28 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Cancer of the Prostate; Neoplasms, Prostate; Prostate Cancer; Prostatic Cancer; Neoplasms, Prostatic; Prostate Neoplasms, Castration-resistant
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASN001: Escalating dose Part A (Experimental): The dose of ASN001 will be based on the assigned study group. The initial dose level of ASN001 will be 50 mg daily. After a safety review, the dose may be escalated for the next group of subjects. Additional dose levels are 100 mg, 200 mg, 300 mg, and 400 mg.
  Interventions: Drug: ASN001: Escalating dose Part A

INTERVENTIONS:
Drug: ASN001: Escalating dose Part A — Androgen inhibitor

SUMMARY:
This study will be conducted in three parts. Part A is a dose-escalation study to determine two safe and tolerable doses of ASN001 for men with metastatic castration resistant prostate cancer. Part A will also characterize the pharmacokinetics and pharmacodynamics of the ASN001 through blood sampling. Subjects in Part B will receive one of two doses identified in Part A to determine which one is more effective, and collect additional pharmacokinetic data. Part C is an extension for subjects completing either Part A or B.

DETAILED DESCRIPTION:
Parts A and B will include a screening period (up to 28 days) and a 12-week treatment period. A subject with no serious adverse drug reactions and who is expected to benefit from continued treatment in the opinion of the investigator will have the opportunity to participate in the long-term extension (Part C). If the subject is not a candidate for or chooses not to participate in the long-term extension (Part C), a post-treatment period of 4 weeks will commence that concludes with an end-of-study visit.

Subjects participating in only Part A or Part B will have approximately 9 study site visits over 18 weeks. Part C will include monthly visits to the study site for 9 months. Thereafter, visits will occur every 3 months. A subject with stable disease or response may continue ASN001 treatment with the approval of the investigator; treatment can continue until a subject experiences an intolerable adverse event (AE) or disease progression, withdraws consent or until termination of the study by the sponsor. At the end of treatment, a post-treatment period of 4 weeks will commence that concludes with an end-of-study visit.

Part B of the study will not be completed as enrollment was halted after Part A (Phase 1)

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed adenocarcinoma of the prostate.
* Ongoing androgen deprivation therapy with a luteinizing hormone-releasing hormone (LHRH) agonist or antagonist, or bilateral orchiectomy and serum testosterone level < 50 ng/dL (< 0.5 ng/mL, < 1.7 nmol/L) at screening
* Metastatic disease documented by computed tomography (CT)/magnetic resonance imaging (MRI) or bone scan.
* Progressive disease despite ongoing androgen deprivation therapy.
* Adequate liver, kidney, and bone marrow function
* Life expectancy of at least 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 at screening
* Patients with prior cytotoxic chemotherapy are eligible to participate if they have been progression free for at least 12 months since the initiation of cytotoxic chemotherapy

Exclusion Criteria:

* Patients with rapidly progressive disease who are candidates for other approved therapies such as docetaxel, abiraterone, and enzalutamide.
* Prior therapy with abiraterone, orteronel, ketoconazole, or any other Cytochrome P450 (CYP) 17 lyase inhibitor; enzalutamide or other experimental androgen receptor antagonist; or experimental immunotherapy agent.
* History of impaired adrenal gland function
* Any investigational treatments for any condition within 4 weeks prior to the start of study treatment.
* Therapy with herbal products known to effect PSA, or estrogen within 30 days prior to the start of study medication
* Known gastrointestinal disease or condition that affects the absorption of ASN001, or difficulty swallowing large capsules.
* Use of systemic glucocorticoid (eg, prednisone, dexamethasone) within 14 days prior to the start of study medication
* Major surgery within 30 days of study medication
* Known brain metastasis
* Previous history of another cancer within 5 years, except completely removed basal or squamous cell skin cancer.
* Serious concurrent medical conditions including: serious heart disease, heart conduction abnormalities, persistent infection, uncontrolled psychiatric illness, liver cirrhosis, chronic liver disease, active or symptomatic viral hepatitis, any other condition that may place the subject at an increased risk or confound the results of the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-01-19 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2017-08-17 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) of ASN001 | First 28 days
  The MTD will be determined by evaluating the number of subjects with treatment related dose limiting toxicity.

SECONDARY OUTCOMES:
Calculate the pharmacokinetic profile of ASN001 | First 29 days
  Pharmacokinetic Parameters
Change in tumor size by CT, MRI or bone scan | 12 weeks
  measure of efficacy
Change in ECOG performance status (score 0 to 5) from baseline as assessed by the investigator | 12 weeks
  Measure of efficacy
Time on treatment | 52 weeks
  Measure of safety, tolerability and preliminary efficacy

OTHER OUTCOMES:
Concentration of serum bone-specific alkaline phosphatase (BAP) | 12 weeks
  To evaluate the effects of ASN001 on the concentration of serum bone-specific alkaline phosphatase (BAP)
The effect of ASN001 on steroid biosynthesis | 52 weeks
  Effects on Luteinizing hormone, follicle stimulating hormone, cortisol, adrenocorticotropic hormone, deoxycorticosterone, corticosterone, dehydroepiandrosterone (DHEA), DHEA sulfate, testosterone and dihydrotestosterone

CONTACTS AND LOCATIONS:
Overall Officials: Niranjan Rao, PhD, Study Director — Asana BioSciences
Locations (6):
- United States (6):
  - UCLA Medical Center, Clark Urology Center, Los Angeles, California
  - Karmanos Cancer Institute, Detroit, Michigan
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Abramson Cancer Center, Hospital of the Univ. of Pennsylvania, Philadelphia, Pennsylvania
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No